CLINICAL TRIAL: NCT04482998
Title: Efficacy of Various Treatments for Acute Acoustic Trauma in the Israeli Defense Force.
Brief Title: Efficacy of Various Treatments for Acute Acoustic Trauma.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Medical Corps, Israel Defense Force (Other)
Responsible Party: Principal Investigator, Yoni Gutkovich, deputy of the head of department for the human performance laboratory, the Israeli naval institute, Haifa., Medical Corps, Israel Defense Force
Other Study IDs: 2131-2020
Record Dates: First submitted 2020-07-19; First posted 2020-07-23 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Acute Acoustic Trauma
Keywords: Hyperbaric Oxygen Therapy; Acute Acoustic Trauma; Steroids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Steroids only - early: treatment was initiated within 7 days of acoustic trauma.
  Interventions: Other: No intervention - retrospective study
- Early combined steroid and hyperbaric oxygen therapy: treatment was initiated within 7 days of acoustic trauma.
  Interventions: Other: No intervention - retrospective study
- Delayed combined steroid and hyperbaric oxygen therapy: treatment was initiated after 7 days of acoustic trauma.
  Interventions: Other: No intervention - retrospective study
- Early sequential steroid followed by HBO therapy: treatment was initiated within 7 days of acoustic trauma.
  Interventions: Other: No intervention - retrospective study
- Delayed sequential steroid followed by HBO therapy: treatment was initiated after 7 days of acoustic trauma.
  Interventions: Other: No intervention - retrospective study
- Hyperbaric oxygen therapy only
  Interventions: Other: No intervention - retrospective study
- No treatment
  Interventions: Other: No intervention - retrospective study
- Steroid only - delayed: treatment was initiated after 7 days of acoustic trauma.
  Interventions: Other: No intervention - retrospective study

INTERVENTIONS:
Other: No intervention - retrospective study — No intervention - retrospective study

SUMMARY:
Acute acoustic trauma is a growing concern in the IDF. there is currently no accepted treatment. The present retrospective study is intended to evaluate the efficacy of different treatment modalities in the IDF between 01/01/2010 and 15/06/2020.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with acute acoustic trauma.
* Hearing exam performed at least 24 hours after acute acoustic trauma.
* There was a reduction of at least 30dB in the 3,000-8,000 Hz frequency range in the first hearing exam performed.

Exclusion Criteria:

* A known hearing impairment prior to acute acoustic trauma.
* Subjects lost from follow up.
* Another diagnosis is more likely than hearing loss due to acute acoustic trauma.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Subjects that served in the IDF and sustained an acute acoustic trauma between 01.01.2010 and 15.06.2020.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Hearing improvement | until 1 year of acoustic trauma.
  dB

SECONDARY OUTCOMES:
Tinnitus | until 1 year of acoustic trauma.
  Qualitative - subjective
Otoacoustic Emissions (OAE) | until 1 year of acoustic trauma.
  dB

CONTACTS AND LOCATIONS:
Locations (1):
- Israeli Navy Medical Institute, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gutkovich YE, Manheim M, Veler R, Geva A, Tal D. Hyperbaric oxygen therapy and corticosteroids as combined treatment for acute acoustic trauma. Eur Arch Otorhinolaryngol. 2025 Jul;282(7):3489-3497. doi: 10.1007/s00405-025-09246-7. Epub 2025 Jan 25. PMID 39863812